CLINICAL TRIAL: NCT03903094
Title: A Retrospective Database Analysis of Anticholinergic Burden Among the Elderly With and Without Overactive Bladder in Australia and South Korea
Brief Title: A Study on Anticholinergic Use: Attribution of Overactive Bladder (OAB) Medications to the Anticholinergic Burden
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Singapore Pte. Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 178-MA-3241
Record Dates: First submitted 2019-03-25; First posted 2019-04-04 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Overactive Bladder (OAB)
Keywords: anticholinergic burden; anticholinergic; overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects With Overactive Bladder Treatment: Subjects who have dispensing records for treatment of overactive bladder will be included
  Interventions: Other: Non-Interventional
- Subjects Without Overactive Bladder Treatment: Subjects who do not have dispensing records for treatment of overactive bladder will be included
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Overview of anticholinergic burden, rather than to evaluate specific drugs

SUMMARY:
Outpatients with at least one dispensing record of any medication will be included in the study. An index date will be assigned to each participant and prescription records for anticholinergics will be used in the study.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one dispensing of any medication between January 22, 2016 and December 31, 2016.

Inclusion Criteria for Korea:

* Have at least one dispensing of any medication between January 1st, 2016 and December 31, 2016.
* Participant was diagnosed with OAB (ICD-10 N32.8, N31.0, N31.1, N31.2, N31.8, N31.9, N32.9, N39.8 and N39.40) at index date.
* Participant did not have dispensing record of an OAB medication during the washout period (6 months prior to the index date).

Exclusion Criteria:

* Participants who do not have a complete year of data availability in the database prior to index date.
* Have record of hospitalization on the index date.

Exclusion Criteria for Korea:

* Participant was hospitalized on the index date.
* Participant did not have an active insurance status during the washout period or on the index date.
* Participant received onabotulinumtoxin A and/or surgical intervention as part of the OAB treatment during the washout period.
* Participant was diagnosed with stress incontinence (ICD-10 N39.3 or equivalent) or had dispensing record of medication for stress incontinence (duloxetine) during the washout period.
* Participant was diagnosed with urinary tract infection (ICD-10 N30.0 and N39.0 or equivalent) during the washout period or on the index date.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Australian and Korean with at least one prescription of any treatment between January 22, 2016 (For Korea: January 1st, 2016) and December 31, 2016 derived from country claims data.
Sampling Method: Non-Probability Sample
Enrollment: 6295279 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Anticholinergic Cognitive Burden (ACB) score | 100 days
  ACB will be calculated based on methodology from Campbell et al (2016). Sum (Drug A #days prescribed X ACB scale score) + (Drug B #days prescribed X ACB scale score) + (Drug X…)/Number of days with any medication prescribed. The cumulative score has a range from 0 to infinity, with higher values indicating a higher cumulative anticholinergic burden of the patient.
Korea Specific: Percentage of Participants With any Listed Anticholinergic Use | 100 days
  This will be calculated as number of participants with any listed anticholinergics use divided by number of participants fulfilling the general eligibility criteria of the study (in each study dataset) multiplied by 100.
Korea Specific: Percentage of Participants With Strong Anticholinergic Use | 100 days
  This will be calculated as number of participants with strong anticholinergics use divided by number of participants fulfilling the general eligibility criteria of the study (in each study dataset) multiplied by 100.
Korea Specific: Number of Anticholinergics Dispensed per Participants | 100 days
  This will be calculated as total number of anticholinergics dispensed divided by number of participants fulfilling the general eligibility criteria of the study (in each study dataset) multiplied by 100.
Korea Specific: Attribution Proportion of OAB medications to total ACB in OAB Cohort | 100 days
  Attribution proportion of OAB medication to total ACB will be calculated as the ratio between the sum over all OAB patients of the ACB scores of each OAB medication multiplied by the number of days supply in the numerator and the sum over all OAB patients of the ACB scores of each antimuscarinic medication multiplied by the number of days supply in the denominator.

SECONDARY OUTCOMES:
Median percentage of ACB score derived from overactive bladder (OAB) treatment(s) in total ACB score | 100 days
  The attribution of antimuscarinics for OAB treatment to entire anticholinergic exposures in OAB patients.

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Global Development, Inc.
Locations (2):
- Site AU61001, Melbourne, Australia
- Site KR82001, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.